CLINICAL TRIAL: NCT01908374
Title: A Randomized, Controlled, Crossover Study to Evaluate the Acute and Subchronic Bioavailability of Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA) From Two Dietary Supplements in Men and Women With Mildly Elevated Triglycerides
Brief Title: Bioavailability of EPA and DHA From Two Dietary Supplements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arctic Nutrition AS (Industry)
Collaborators: BioFortis (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PRV-1302
Record Dates: First submitted 2013-07-19; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Hypertriglyceridemia
Keywords: Active-placebo controlled double blind cross over
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHA-rich fish oil (Active Comparator): DHA-rich fish oil versus Phospholipid-rich fish oil Fish oil in triglyceride form (12 capsules/d providing 575 mg/d EPA; 1843 mg/d DHA; 259 mg/d n-3 DPA)
  Interventions: Dietary Supplement: DHA-rich fish oil versus Phospholipid-rich fish oil
- Phospholipid-rich fish oil (Experimental): DHA-rich fish oil versus Phospholipid-rich fish oil Fish roe high in EPA/DHA phospholipids [(12 capsules/d providing 628 mg/d EPA; 1810 mg/d DHA; 137 mg/d n-3 docosapentaenoic acid (DPA)]
  Interventions: Dietary Supplement: DHA-rich fish oil versus Phospholipid-rich fish oil

INTERVENTIONS:
Dietary Supplement: DHA-rich fish oil versus Phospholipid-rich fish oil — This randomized, controlled crossover study will include four treatment visits (visits 2, 3, 4, and 5; days 0, 14, 42, and 56). Subjects will be randomly assigned, by sex and age, to their first treatment study product (active or control), which will be administered with a standardized low-choline, DHA-, EPA- free breakfast meal at t = 0 h. Subjects will consume placebo or phospholipid-rich fish oil for two weeks, washed out for 4 weeks, then treatments switched. Blood samples will be obtained for acute measurements on visits 2 and 4, via an indwelling venous catheter or venipuncture at t = 1, 2, 4, 6, 8, 10, and 12 h ± 5 min, to determine plasma fatty acid profile. Chronic fatty acid measurements will be determined after 2 weeks on visits 3 and 5.
  Other Names: MOPL(TM)30; Marine Omega-3 Phospholipids; Herring Caviar Phospholipids

SUMMARY:
The primary objective of this study is to test the effects of two different fish oil products containing DHA and EPA by comparing the omega-3 fatty acid levels in the blood.

DETAILED DESCRIPTION:
The objective of this study is to evaluate and compare the acute and sub-chronic (2 week) bioavailability of EPA and DHA from two marine oil supplements consumed with a meal in men and women with mildly elevated triglycerides. The supplements provide similar amounts of EPA + DHA esterified as either triglycerides; or esterified as phospholipids and triglycerides.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 18-59 years of age, inclusive.
2. Subject has a body mass index (BMI) of ≥18.50 and ≤29.99 kg/m2 at visit 1b (day -7).
3. Subject has a score of 7 to 10 on the Vein Access Scale at visit 1b (day -7; Appendix 3).
4. Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine laboratory test results.
5. Subject has a fasting TG 100-249 mg/dL at visit 1b (day -7). One venous retest allowed if ≥250 mg/dL.
6. Subject is willing to refrain from consumption of all fish/seafood (including shellfish), foods rich in choline, fatty acid-containing foods and supplements, and/or EPA-, DHA-containing foods and supplements (≤1.0 g/d ) 14 d prior to visit 2 (day 0) and throughout the study (Appendix 1).
7. Subject is willing to limit alcohol consumption to no more than 1 drink/d following visit 1b (day -7) and throughout the study.
8. Subject has no plans to change smoking habits during the study period and agrees to abstain from tobacco products for at least 1 h prior to and throughout the duration of the clinic visits [visits 1b, 3 and 5 (days -7, 14 and 56) for up to 2 h; and visits 2 and 4 (days 0 and 42) for up to 14 h].
9. Subject is willing to comply with fecal collection procedures.
10. Subject is willing to maintain habitual diet (with the exception of foods to be restricted), physical activity patterns, and body weight throughout the trial.
11. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subject is male or female, 18-59 years of age, inclusive.
2. Subject has a body mass index (BMI) of ≥18.50 and ≤29.99 kg/m2 at visit 1b (day -7).
3. Subject has a score of 7 to 10 on the Vein Access Scale at visit 1b (day -7; Appendix 3).
4. Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine laboratory test results.
5. Subject has a fasting TG 100-249 mg/dL at visit 1b (day -7). One venous retest allowed if ≥250 mg/dL.
6. Subject is willing to refrain from consumption of all fish/seafood (including shellfish), foods rich in choline, fatty acid-containing foods and supplements, and/or EPA-, DHA-containing foods and supplements (≤1.0 g/d ) 14 d prior to visit 2 (day 0) and throughout the study (Appendix 1).
7. Subject is willing to limit alcohol consumption to no more than 1 drink/d following visit 1b (day -7) and throughout the study.
8. Subject has no plans to change smoking habits during the study period and agrees to abstain from tobacco products for at least 1 h prior to and throughout the duration of the clinic visits [visits 1b, 3 and 5 (days -7, 14 and 56) for up to 2 h; and visits 2 and 4 (days 0 and 42) for up to 14 h].
9. Subject is willing to comply with fecal collection procedures.
10. Subject is willing to maintain habitual diet (with the exception of foods to be restricted), physical activity patterns, and body weight throughout the trial.
11. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve for plasma phosphatidylcholine omega-3 fatty acids | pre-dose, 1, 2, 4, 6, 8, 10, 12 hours post-dose
  The primary outcome variable will be the net incremental area under the curve (niAUC) for plasma phosphatidylcholine (PC) EPA + DHA from pre-meal (t = -0.5 h pre-dose) to 12 h post-dose (niAUC 0-12 h post-dose) measured at visits 2 and 4 (analyzed with and without normalization to the intake of EPA+DHA in each group).

SECONDARY OUTCOMES:
Maximum concentration and Time to maximum concentration for plasma omega-3 phosphatidylcholine fatty acids | pre-dose, 1, 2, 4, 6, 8, 10, 12 hours post-dose
  The maximal concentration (Cmax) and time to Cmax (Tmax) for plasma PC EPA + DHA, EPA, DHA, DPA, and EPA + DHA + DPA (analyzed with and without normalization to the intake of EPA, DHA, DPA, and EPA+DHA+DPA in each group) from pre-meal to 12 h post-dose at visits 2 and 4.
Area under the curve for plasma phosphatidylcholine omega-3 fatty acids Part 2 | pre-dose, 1, 2, 4, 6, 8, 10, 12 hours post-dose
  The niAUC for plasma PC EPA; PC DHA; PC DPA; PC EPA + DHA + DPA from pre-meal (t = -0.5 h pre-dose) to 12 h post-dose (niAUC0-12 h) at visits 2 and 4 (analyzed with and without normalization to the intake of EPA, DHA, DPA, and EPA+DHA+DPA in each group).
Plasma sphingomyelin and total plasma phosphatidylcholine | pre-dose, 0, 1, 2, 4, 6, 8, 10, 12 hours post-dose
  Plasma sphingomyelin and total plasma PC at visits 2, 3, 4, and 5
Fasting plasma lipoprotein lipids | pre-dose
  Percent changes from baseline (average of values at visits 1 and 2) to the end of each treatment period (visits 3,4,5) in the following fasting lipoprotein lipids: high-density lipoprotein cholesterol (HDL-C), non-HDL-C, low-density lipoprotein cholesterol (LDL-C), total cholesterol (TC), triglycerides, and high sensitivity C reactive protein (hs-CRP).
Gastrointestinal (GI) Tolerability Questionnaire | 0, 12 hours post-dose
  Ratings from the GI Tolerability Questionnaire
Product Acceptability Questionnaire | 0, 12 hours post-dose
  Ratings from the Product Acceptability Questionnaire
Adverse Events (AE) | pre-treatment, 0, 12 hours post-dose
  AE assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, Ph. D, Study Director — BioFortis; Kathleen Kelley, M.D., Principal Investigator — BioFortis
Locations (1):
- Biofortis, Addison, Illinois, United States

REFERENCES:
- [Background] Davidson MH, Maki KC, Bays H, Carter R, Ballantyne CM. Effects of prescription omega-3-acid ethyl esters on lipoprotein particle concentrations, apolipoproteins AI and CIII, and lipoprotein-associated phospholipase A(2) mass in statin-treated subjects with hypertriglyceridemia. J Clin Lipidol. 2009 Oct;3(5):332-40. doi: 10.1016/j.jacl.2009.08.001. Epub 2009 Aug 31. PMID 21291831
- [Background] Davidson MH, Johnson J, Rooney MW, Kyle ML, Kling DF. A novel omega-3 free fatty acid formulation has dramatically improved bioavailability during a low-fat diet compared with omega-3-acid ethyl esters: the ECLIPSE (Epanova((R)) compared to Lovaza((R)) in a pharmacokinetic single-dose evaluation) study. J Clin Lipidol. 2012 Nov-Dec;6(6):573-84. doi: 10.1016/j.jacl.2012.01.002. Epub 2012 Jan 24. PMID 23312053
- [Background] Grimsgaard S, Bonaa KH, Hansen JB, Nordoy A. Highly purified eicosapentaenoic acid and docosahexaenoic acid in humans have similar triacylglycerol-lowering effects but divergent effects on serum fatty acids. Am J Clin Nutr. 1997 Sep;66(3):649-59. doi: 10.1093/ajcn/66.3.649. PMID 9280188
- [Background] Maki KC, Reeves MS, Farmer M, Griinari M, Berge K, Vik H, Hubacher R, Rains TM. Krill oil supplementation increases plasma concentrations of eicosapentaenoic and docosahexaenoic acids in overweight and obese men and women. Nutr Res. 2009 Sep;29(9):609-15. doi: 10.1016/j.nutres.2009.09.004. PMID 19854375
- [Background] Miller M, Stone NJ, Ballantyne C, Bittner V, Criqui MH, Ginsberg HN, Goldberg AC, Howard WJ, Jacobson MS, Kris-Etherton PM, Lennie TA, Levi M, Mazzone T, Pennathur S; American Heart Association Clinical Lipidology, Thrombosis, and Prevention Committee of the Council on Nutrition, Physical Activity, and Metabolism; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease. Triglycerides and cardiovascular disease: a scientific statement from the American Heart Association. Circulation. 2011 May 24;123(20):2292-333. doi: 10.1161/CIR.0b013e3182160726. Epub 2011 Apr 18. No abstract available. PMID 21502576
- [Background] Mori TA, Burke V, Puddey IB, Watts GF, O'Neal DN, Best JD, Beilin LJ. Purified eicosapentaenoic and docosahexaenoic acids have differential effects on serum lipids and lipoproteins, LDL particle size, glucose, and insulin in mildly hyperlipidemic men. Am J Clin Nutr. 2000 May;71(5):1085-94. doi: 10.1093/ajcn/71.5.1085. PMID 10799369
- [Background] Schuchardt JP, Schneider I, Meyer H, Neubronner J, von Schacky C, Hahn A. Incorporation of EPA and DHA into plasma phospholipids in response to different omega-3 fatty acid formulations--a comparative bioavailability study of fish oil vs. krill oil. Lipids Health Dis. 2011 Aug 22;10:145. doi: 10.1186/1476-511X-10-145. PMID 21854650
- [Background] Ulven SM, Kirkhus B, Lamglait A, Basu S, Elind E, Haider T, Berge K, Vik H, Pedersen JI. Metabolic effects of krill oil are essentially similar to those of fish oil but at lower dose of EPA and DHA, in healthy volunteers. Lipids. 2011 Jan;46(1):37-46. doi: 10.1007/s11745-010-3490-4. Epub 2010 Nov 2. PMID 21042875